CLINICAL TRIAL: NCT06907511
Title: A Phase 1/2, Parallel-group, Randomized, Modified Double-blind, Placebo-controlled, Multi-center, Dose Ranging Study to Evaluate the Safety and Immunogenicity of a Second Generation Structurally Designed Pandemic Influenza H5 HA mRNA Vaccine in Healthy Adults Aged 18 Years and Older
Brief Title: Study to Evaluate the Safety and the Immunogenicity of a Second Generation Structurally Designed mRNA Vaccine Candidate Against Pandemic Influenza H5 HA Strain in Healthy Adult Participants Aged 18 Years and Older
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VBS00002; U1111-1314-5493 (Other: WHO ICTRP)
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pandemic Influenza Immunization; Healthy Volunteers
Keywords: Pandemic Flu H5 Vaccination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind (participants; sites, except for those preparing/administering study intervention; and Sponsor will be blinded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: Pandemic flu H5 HA mRNA SD2 vaccine (Low dose) (Experimental): Participants will receive two injections of low dose pandemic flu H5 HA mRNA SD2 vaccine
  Extension Phase:
  Additional participants will receive two injections 21 days apart of pandemic flu H5 HA mRNA SD2 vaccine at low dose
  Interventions: Biological: Pandemic flu H5 HA mRNA SD2 vaccine
- Group 2: Pandemic flu H5 HA mRNA SD2 vaccine (Medium dose) (Experimental): Participants will receive two injections of medium dose pandemic flu H5 HA mRNA SD2 vaccine
  Interventions: Biological: Pandemic flu H5 HA mRNA SD2 vaccine
- Group 3: Pandemic flu H5 HA mRNA SD2 vaccine (High dose) (Experimental): Participants will receive two injections of high dose pandemic flu H5 HA mRNA SD2 vaccine
  Interventions: Biological: Pandemic flu H5 HA mRNA SD2 vaccine
- Group 4: Placebo (Placebo Comparator): Participants will receive two injections of placebo
  Extension Phase:
  Additional participants will receive two injections 21 days apart of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Pandemic flu H5 HA mRNA SD2 vaccine — Pharmaceutical Form:
  Suspension in a vial
  Route of Administration:
  Intramuscular injection
  Arms: Group 1: Pandemic flu H5 HA mRNA SD2 vaccine (Low dose); Group 2: Pandemic flu H5 HA mRNA SD2 vaccine (Medium dose); Group 3: Pandemic flu H5 HA mRNA SD2 vaccine (High dose)
Other: Placebo — Pharmaceutical Form:
  Liquid solution in a vial
  Route of Administration:
  Intramuscular injection
  Arms: Group 4: Placebo

SUMMARY:
The purpose of this phase 1/2 study is to investigate the safety and immunogenicity of different doses (high, medium and low) of a second generation structurally designed (SD2) H5 messenger ribonucleic acid (mRNA) vaccine against pandemic H5 influenza virus (pandemic flu H5 hemagglutinin (HA) mRNA SD2) in healthy younger and older adults.

The study will aim to identify the appropriate dose for further clinical development of a potential pandemic response vaccine.

The study also includes an extension phase for one of the 3 dose levels of the pandemic flu H5 HA mRNA SD2 vaccine to collect additional safety and the immunogenicity data for this specific dose of the vaccine. During this Extension Phase, an additional 480 participants will be randomized according to a 1:1 ratio and stratified by age (≥ 18 to < 65 years and ≥ 65 years) to receive either the low dose of the pandemic flu H5 HA mRNA DS2 vaccine (Group 1) or placebo (Group 4). This extension will enhance the safety database and improve precision of the immunogenicity results for the selected dose while preserving the original study design integrity.

The study duration per participant will be approximately 13 months. There will be two injections of placebo or pandemic flu H5 mRNA vaccine 21 days apart at high, medium and low doses.

Study visits/contact include: 7 study visits and 1 telephone call. Vaccination visits (including blood samples) will occur at Day 01 and Day 22. Short-term follow-up visits (including blood samples) will occur 8 and 21 days after each injection. Participants will be also followed up (including blood samples) at 3 and 6 months after 2nd injection, and at 12 months after 2nd injection for safety.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older on the day of inclusion
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, or surgically sterile.

OR

• Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to each study intervention administration until at least 12 weeks after the last study intervention administration

* A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) within 8 hours before the first dose of study intervention

Exclusion Criteria:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the study intervention components (eg, polyethylene glycol, polysorbate); history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances; any allergic reaction (eg, anaphylaxis) after administration of an mRNA vaccine
* Previous history of myocarditis, pericarditis, and/or myopericarditis
* Known history of previous episodes of Guillain-Barré Syndrome (GBS), neuritis (including Bell's palsy), convulsions , encephalitis, transverse myelitis, and vasculitis
* Participants with an electrocardiogram that is consistent with possible myocarditis or pericarditis or, in the opinion of the investigator, demonstrates clinically relevant abnormalities that may affect participant safety or study results
* Self-reported thrombocytopenia, contraindicating IM injection based on investigator's judgment
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM injection based on investigator's judgment
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness / infection (according to investigator's judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of study intervention. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Alcohol, prescription drug, or substance abuse that, in the opinion of the investigator, might interfere with the study conduct or completion
* Participant who had acute infectious symptoms or a positive severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) reverse transcriptase polymerase chain reaction (RT PCR) or antigen test in the past 10 days prior to the first visit (V)01
* Receipt of any vaccine other than an mRNA vaccine in the 4 weeks preceding study intervention administration or planned receipt of any vaccine other than an mRNA vaccine in the 3 weeks following the second dose of the study intervention
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Receipt of any mRNA vaccine/product in the 2 months preceding study intervention administration or planned receipt of any mRNA vaccine in the 2 months after the second dose of the study intervention
* Participation at the time of study enrollment (or in the 4 weeks preceding study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Previous history of participation in an H5 influenza A vaccine study. This includes any influenza subtypes that contain H5 such as H5N1, H5N8, or H5N6

Note: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Presence of immediate adverse events (AEs) | Within 30 minutes after each/any injection
  Number of participants with immediate AEs
Presence of solicited injection site reactions | Through 7 days after each/any injection
  Number of participants with solicited injection site reactions
Presence of solicited systemic reactions | Through 7 days after each/any injection
  Number of participants with solicited systemic reactions
Presence of unsolicited AEs | Through 21 days after the first injection through 28 days after the second injection
  Number of participants with unsolicited AEs
Presence of medically attended adverse events (MAAEs) | Through 180 days after the last injection
  Number of participants with MAAEs
Presence of adverse events of special interest (AESIs) | Throughout the study, approximately 13 months
  Number of participants with AESIs
Presence of serious adverse events (SAEs) | Throughout the study, approximately 13 months
  Number of participants with SAEs
Presence of out-of-range biological test results (including shift from baseline values) | Through a maximum of 8 days after each injection
  Number of participants with out-of-range biological test results

SECONDARY OUTCOMES:
Geometric mean titers (GMTs) of antibodies (Abs) against investigational pandemic flu H5 HA mRNA SD2 vaccine | Day 01, Day 22, Day 43, Day 112 and Day 202
  Ab titer measured by hemagglutination inhibition (HAI) assay
Individual HA titer ratio | Day22/Day01, Day43/Day01, Day112/Day01, and Day202/Day01
  Geometric mean ratio (GMR) HAI titers ratio
Seroconversion HAI Titer | Day 01, Day 22 and Day 43
  Percentage of participants with seroconversion
  Seroconversion is defined by:
  HAI titer < 10 [1/dilution (dil)] on Day 01 and post-injection titer ≥ 40 [1/dil] on Day 22 or Day 43; or defined as HAI titer ≥ 10 [1/dil] on D01 and a ≥ 4-fold increase in titer [1/dil]) on Day 22 or Day 43
HAI titer ≥ 40 (1/dil) | Day 01, Day 22, Day 43, Day 112, and Day 202
  Percentage of participants with HAI titer ≥ 40 (1/dil)
Detectable HAI titer ≥ 10 (1/dil) | Day 01, Day 22, Day 43, Day 112, and Day 202
  Percentage of participants with HAI titer ≥ 10 (1/dil)
GMTs of Abs against investigational pandemic flu H5 HA mRNA SD2 vaccine | Day 01, Day 22, Day 43, Day 112 and Day 202
  Ab titer measured by seroneutralization (SN) test
Individual SN titer ratio | Day 22/Day 02, Day 43/Day 01, Day 112/Day 01 and Day 202/Day 01
  GMR SN titers ratio
SN titer ≥ 20 (1/dil) | Day 01, Day 22, Day 43, Day 112 and Day 202
  Percentage of participants with SN titer ≥ 20 (1/dil)
SN titer ≥ 40 (1/dil) | Day 01, Day 22, Day 43, Day 112 and Day 202
  Percentage of participants with SN titer ≥ 40 (1/dil)
SN titer ≥ 80 (1/dil) | Day 01, Day 22, Day 43, Day 112 and Day 202
  Percentage of participants with SN titer ≥ 80 (1/dil)
Detectable SN titer ≥ 10 (1/dil) | Day 01, Day 22, Day 43, Day 112, and Day 202
  Percentage of participants with SN titer ≥ 10 (1/dil)
2-fold and 4-fold rise in SN titer | Day 22 and Day 43
  Percentage of participants with fold increase in SN Ab titer [post-vaccination / pre- vaccination] ≥ 2 and ≥ 4 on D22 and D43

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Velocity Clinical Research - San Diego- Site Number : 8400013, La Mesa, California
  - Accel Research Sites Network - DeLand Clinical Research Unit- Site Number : 8400002, DeLand, Florida
  - Accel Research Sites - Lakeland Clinical Research Unit- Site Number : 8400006, Lakeland, Florida
  - Accel Research Sites - St. Petersburg - Largo- Site Number : 8400004, Largo, Florida
  - Accel Research Site - NeuroStudies.net, LLC - ERN - PPDS- Site Number : 8400003, Decatur, Georgia
  - QUEST Research Institute- Site Number : 8400014, Bingham Farms, Michigan
  - Velocity Clinical Research - Norfolk- Site Number : 8400015, Norfolk, Nebraska
  - Velocity Clinical Research - Omaha- Site Number : 8400012, Omaha, Nebraska
  - Velocity Clinical Research - Springdale- Site Number : 8400010, Cincinnati, Ohio
  - Coastal Carolina Research Center- Site Number : 8400001, North Charleston, South Carolina
  - Olympus Clinical Research - Sugar Land- Site Number : 8400009, Sugar Land, Texas
  - Velocity Clinical Research - Salt Lake City- Site Number : 8400011, West Jordan, Utah
  - Charlottesville Medical Research- Site Number : 8400005, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org.

REFERENCES:
- See also: VBS00002 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26645&tenant=MT_SNY_9011